CLINICAL TRIAL: NCT00947284
Title: Effect of Kappa Opioid Agonist-Antagonists in the Heat/Capsaicin Sensitization Model
Brief Title: Effect of Nalbuphine and Naloxone on Experimentally Induced Skin Sensitivity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Experimental pain model didn't work as anticipated.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NIH/NIDCR R01 DE018526-2; 5R01DE018526-02 (NIH)
Record Dates: First submitted 2009-07-01; First posted 2009-07-28 (Estimated); Results first posted 2013-10-23 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — Nalbuphine; Naloxone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Women (Experimental): Both arms of this study will receive identical interventions. The only difference will be the sex of the participants in each study arm.
  Interventions: Drug: nalbuphine plus naloxone; Drug: nalbuphine plus saline; Drug: naloxone plus saline
- Men (Experimental): Both arms of this study will receive identical interventions. The only difference will be the sex of the participants in each study arm
  Interventions: Drug: nalbuphine plus naloxone; Drug: nalbuphine plus saline; Drug: naloxone plus saline

INTERVENTIONS:
Drug: nalbuphine plus naloxone — single dose administered intravenously
  Other Names: Nubain; Narcan
Drug: nalbuphine plus saline — single dose administered intravenously
  Other Names: Nubain
Drug: naloxone plus saline — single dose administered intravenously
  Other Names: Narcan

SUMMARY:
In previous clinical studies of post-surgical pain the investigators found that nalbuphine (Nubain), a narcotic pain killer, relieves pain more effectively when combined with low-dose naloxone (Narcan), a drug that is used to treat narcotic overdose. This finding was particularly true in men. The purpose of this study is to find out if nalbuphine combined with naloxone is more effective in relieving experimentally produced pain than either drug alone. A second reason for this study is to find out if study medications work more effectively in women or in men. Subjects will come to the University of California at San Francisco (UCSF) Clinical Research Center (CRC) for 4 study visits. The first visit will be a 2-hour screening to assess the subject for study eligibility. During the other three visits, the investigators will use a thermal stimulating device to produce temporary, non-injurious skin sensitivity that subjects will feel as painful. Changes in pain will be measured following the intravenous (i.v.) administration of study drugs. Three drug combinations will be administered, a different one each visit: 1) nalbuphine 5 mg and naloxone 0.4 mg , 2) naloxone 0.4 mg and saline (an inactive solution), nalbuphine 5 mg and saline. These drug combinations will be administered in random order; all subjects will receive all three combinations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 40
* In stable health
* Speak, read, understand English language
* If female, must be non-lactating and not pregnant

Exclusion Criteria:

* Heat pain detection thresholds above 47 ºC/116.6 ºF
* Inability to develop secondary hyperalgesia from the heat and capsaicin stimulation performed at the screening visit
* Serious psychiatric psychopathology (psychotic disorder, substance abuse)
* Tattoos in the area of measurements
* Allergy to study drugs (nalbuphine, naloxone, or capsaicin)
* Current or recent use opioids

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon D Levine, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment details unavailable due to death of investigator
Pre-assignment Details: Pre-assignment details unavailable due to death of investigator
Groups:
- Women-all Three Combinations; Men-all Three Combinations: the investigators will use a thermal stimulating device to produce temporary, non-injurious skin sensitivity that subjects will feel as painful. Changes in pain will be measured following the intravenous (i.v.) administration of study drugs. Three drug combinations will be administered, a different one each visit: 1) nalbuphine 5 mg and naloxone 0.4 mg , 2) naloxone 0.4 mg and saline (an inactive solution), nalbuphine 5 mg and saline. These drug combinations will be administered in random order; all subjects will receive all three combinations.
Period: Overall Study
Arm/Group | Women-all Three Combinations | Men-all Three Combinations
Started | 0 | 3
Completed | 0 | 0
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Arm/Group | Men-all Three Combinations
Number analyzed (Participants) | 3
Age, Customized [Number; unit: Participants] — Demographic data not available due to death of investigator; co-investigators searched the computer of the deceased investigator and cannot find additional data
  Participants
    Unknown | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Skin Sensitivity as Measured by a Visual Analog Scale
Description: Participants would have been asked to rate the level of pain on a scale from 0 (no pain) to 10 (worst pain imaginable).
Time Frame: Prior to drug administration and 20 minutes, 70 minutes and 2 hours after each drug administration
Population: The planned model of skin irritation could not be reproduced on 3 enrolled participants, thus the investigator did not obtain outcome data.
Arm/Group | Men-all Three Combinations
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 day
Description: The lead investigator passed away and co-investigators could not find adverse event data on his computer. The experimental model for skin sensitivity did not work in the first 3 participants, and the study was terminated without collecting outcomes data.
Arm/Group | Men-all Three Combinations
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The lead investigator passed away and co-investigators could not find complete data on his computer. The experimental model for skin sensitivity did not work in the first 3 participants, and the study was terminated without collecting outcomes data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes